## VillageWhere:

# Innovative Mobile Technology for Youth with Conduct Disorder and Their Parents Informed Consent Forms

Behavioral Health Research Collective IRB Protocol Number: 030

National Clinical Trial (NCT) Identified Number: NCT03065517

Principal Investigators: Linda Dimeff, PhD & Cindy Schaeffer, PhD

**Sponsor: Evidence-Based Practice Institute, Inc.** 

Grant Title: Using Mobile Technology to Enhance MST | Grant Number: R44MH097349

**Funded by: National Institute of Mental Health** 

Version Number: 3 | 10 November 2019

## iKinnect Clinical Trial

## Evidence-Based Practice Institute, LLC CONSENT TO PARTICIPATE IN RESEARCH – Parent/Guardian & Youth Version

**TITLE:** Developing Mobile Technology to Enhance Multisystemic Therapy (MST)

Outcomes

SPONSOR & National Institute of Mental Health

PROTOCOL NUMBER: R44MH097349-A1

PRINCIPAL Linda Dimeff, PhD INVESTIGATORS: (206) 384-7371

Cindy Schaeffer, PhD

(410) 706-6855

SITE: Evidence-Based Practice Institute, LLC

3303 South Irving Street Seattle, Washington 98144

**United States** 

OTHER STUDY-RELATED Julie Chung

PHONE NUMBER: Study Coordinator

(206) 717-5666

## This consent form contains important information to help you decide whether to participate in a research study.

- > Being in a study is voluntary your choice.
- If you join this study, you can still stop at any time.
- No one can promise that a study will help you.
- Do not join this study unless all of your questions are answered.

## After reading and discussing the information in this consent form you should know:

- Why this research study is being done;
- What will happen during the study;
- Any possible benefits to you;
- The possible risks to you;
- Other options you could choose instead of being in this study;
- How your personal health information will be treated during the study and after the study is over;
- Whether being in this study could involve any cost to you; and
- What to do if you have problems or questions about this study.

## Please read this consent form carefully.

## A. PURPOSE & BACKGROUND

We have developed iKinnect, a new mobile app for teens who have behaviors like skipping school, physical fights, illegal behaviors, and arrests and their parents/guardians. iKinnect is designed to give teens rewards (like Google Play/Apple Store credit) for positive behavior, help parents/guardians and teens work together to meet behavior goals, and monitor teen activities and whereabouts. Right now, we are looking for parents/guardians and teens to use the app for 12 weeks (3 months) in real life and tell us their likes and dislikes as they use it. We will also ask that parents/guardians and teens complete phone interviews and online surveys at the start of the study (baseline) and at 4, 8, and 12 weeks.

You and your teen are being asked to volunteer for this research study. Your participation is completely voluntary (your choice). You do not have to be in this study if you do not want to. Parents/Guardians and teens are required to participate together as a pair. This means that both you and your teen must agree to participate in the study in order to enroll in it. Parents/Guardians and teens will participate together and pairs will be randomly assigned (like flipping a coin) to use either the iKinnect app or another app, called Life360, on your Android or Apple smartphones. All study interviews and surveys will be completed independently (on your own). We will want to talk with you and your teen about your views and opinions about how the app you were assigned to use is working for your family, what you like and dislike, and your suggestions for how to make it better. We will also ask about and evaluate the app's helpfulness/usefulness, how often you and your teen use the app, barriers you might experience to using the app, parenting practices, life stress, clarity of expectations, youth delinquent/prosocial behaviors, and motivation.

Finally, if you and your teen are assigned to use the iKinnect app, we will ask your permission to talk with your service provider (case manager, therapist, etc.) at 8 weeks. We will ask your provider their opinions about your and your teen's use of the app, and whether they believe the app was helpful to youth progress.

## **B. STUDY PROCEDURES**

If you agree to be in this study, the following will happen:

- 1. You and your teen will be randomly assigned (like flipping a coin) as a pair to use either the iKinnect app or the Life360 app on your Android or Apple smartphones.
- 2. We will give you and your teen a link to the iKinnect mobile app or another app used in the study. We will then ask that you each install the app on your Android or Apple smartphones and set it up. We are here to help with this process if you need.
- 3. You will be asked to use the app for 12 weeks. You will not be required to use any particular feature of the app if there is a specific reason why you and/or your teen prefer not to.
- 4. If you are assigned to use the iKinnect app, the research team will be able to access the information collected through your and your teen's use of the app. iKinnect data that we collect will be coded with your study ID number and combined with the other participants' data. We will use this information to determine how iKinnect is being used by the parents/guardians and teens in this study. You will not be asked about this information during the study interview or surveys.
- 5. If you are assigned to use the Life360 app, you will be required to provide the following permissions in order for it to work properly: 1) location; 2) phone permission to allow Life360 to connect your phone to a live representative and authenticate that you are the one calling them if you choose to use that feature; and 3) network to allow Life360 to send and receive location information to and from family members on your private map. Other information regarding their terms of use, privacy policy, and data retention policies can be found in your app store or on the Life360 website.
- 6. You and your teen will each be asked to complete 4 study assessments over your 12 weeks of being in the study. These assessments will take place at the start of your participation (also called

"baseline") and during weeks 4, 8, and 12. Each assessment will include an interview and a brief set of surveys online. We expect no interview to last longer than 30 minutes and the surveys no longer than 30 minutes. Each assessment will last about 1 hour total. The assessments will be scheduled at a time that is most convenient for you and your teen. We recommend ensuring you are in a quiet, private place during the assessments. We will want to talk with you and your teen about your views and opinions on how the app is working for your family, what you like and dislike, and your suggestions for how to make it better. We will also ask about and evaluate the app's helpfulness/usefulness, how often you and your teen use the app, barriers you might experience to using the app, parenting practices, life stress, clarity of expectations, youth delinquent/prosocial behaviors, and motivation.

- 7. You and your teen will each receive compensation for the study assessments you complete and can earn bonuses for completing at least 3 (Bonus 1) and all 4 (Bonus 2) of the assessments. Parents/Guardians can earn up to \$240 and teens can earn up to \$140 for completing this study.
- 8. You and your teen's names will not be associated with the answers you provide during the interviews or on surveys. You have the right to not answer a question or withdraw from the study for any reason at any time if you choose, without penalty. You may contact Dr. Dimeff or Dr. Schaeffer at any time if you have any concerns or are feeling discomfort due to study participation.

#### C. RISKS/DISCOMFORTS

There are seven kinds of potential risks to you and/or your teen for participating in this study:

1. Potential embarrassment of sharing your opinions (likes and dislikes) of the app with us in an interview and/or feeling possible distress when answering survey questions about teen's functioning and parenting behaviors.

## To reduce the risk of embarrassment and/or distress of sharing your opinions and other study data with us:

- During the study interviews, we will talk only about the app itself and how teens, parents/guardians, and service providers might use it; discussions about personal or private matters will not be allowed.
- If at any time you and/or your teen feels uncomfortable or embarrassed, you and/or your teen are encouraged to tell us right away.
- If you would like, we will tell the investigators of you/your teen's concerns, and she will contact you to talk about how best to address your concerns.
- To lessen the anxiety that assessment procedures can cause, we have purposely designed the
  procedure to allow you to complete the assessments in the comfort of your own home. We are
  also available to answer any questions you may have or provide any assistance you might need
  during the assessments.
- You are free to stop your participation in the study at any time or refuse to answer any question you are uncomfortable answering.
- 2. Possibility of experiencing distress if you and your teen disagree about how the app should be used.

## To reduce the possibility of you or your teen experiencing distress if you disagree about how the app should be used:

- Research staff, including staff who are clinical psychologists, will be available to talk with you if this occurs and you would like to speak with someone about it.
- If you or your teen's distress level is high, you, your teen, or a research staff member can inform your service provider about the distress and your provider can help you.

- You are free to withdraw from the study at any time if you find that participation is too distressing.
- 3. Potential embarrassment when using the app in a public place or when around people who you may know or who may not know you are in a research study.

To reduce the risk of embarrassment when using the app in a public place or when around people who you may know or who may not know you are participating in a research study:

- You and your teen are encouraged to only use the app when it feels comfortable to do so.
- We will never require you or your teen to use the app in a place or at a time when you do not want to use it.
- The server that houses the app is as resistant to hacking as possible; the protections for the server are similar to those used in banking or other commercial websites. This will help protect your information stored in the app, such as if the app server were "hacked" or if you or your teen were to lose your phone.
- As an added protection, all app-generated information will be stored on the server without your name. In addition, the app will only store data on the server, not on the phone itself.
- Using the app requires a login, and you can log out of the app at any time.
- Finally, as an added safeguard, we recommend you and your teen password-protect your smartphones (such as using a pin to unlock the phone) while you are in this study.
- 4. Possibility of incurring data charges while using the app.

## To avoid the possibility of incurring data charges while using the app:

- Check with your smartphone's data provider to ensure you know how much data you are allowed to use each billing period without incurring extra charges.
- Use the app only when on a Wi-Fi connection.
- If needed, log out of the app and only log back in when you are comfortable doing so.
- 5. Possible loss of confidentiality and security of your data.

To minimize risks to confidentiality associated with management and storage of data, including identification of participants who took part in this study or information collected about you and your teen while using the app, we will:

- Train and supervise research staff to ensure strict compliance with the data protection plan.
- You and/or your teen's answers during the interviews and on the surveys will be stored on a secure, password-protected drive accessible only to research staff.
- Your and your teen's responses will be stored using a study ID number and the last four digits of your mobile device number. The list linking you and/or your teen's name to the ID assigned to your information will be maintained in a separate, secured location, also password protected and accessible only to the research staff, and will be destroyed within three years from the date of collection.
- The information we collect from you and your teen will be associated only with your study ID
  number and the last four digits of your mobile device number, not your name, so nobody can
  identify it as yours. This is called "de-identified data." De-identified data will be kept indefinitely
  on the secure drive.
- 6. You or your teen could feel coerced (pressured) to participate.

To minimize the risk that you or your teen will feel pressure or coercion to participate:

- You are under no obligation to participate in the study at all. You may stop your participation in the study at any time.
- To ensure that participation is indeed completely voluntary, we have informed your agency staff, including your service provider, on multiple occasions that participation in this study is and must remain completely voluntary (your choice).
- We will ask you and your teen separately for consent/assent to participate and inform each of you independently that being in the study is completely voluntary.
- You and your teen may refuse participation in any part of the study. You and your teen may also discontinue your participation in this study at any time, without in any way jeopardizing your treatment or legal status.
- 7. The final risk involves privacy and the protection of your data.

## To help us protect your and your teen's privacy and data we collect during the study:

We have obtained a Certificate of Confidentiality from the National Institutes of Health. This Certificate helps protect your identifiable research information from forced or compelled disclosure. A Certificate of Confidentiality allows the investigator and others who have access to research records to refuse to disclose identifying information on research participants in civil, criminal, administrative, legislative, or other proceedings, whether federal, state, or local. The researchers will use the Certificate to resist any demands for information that would identify you. Certificates of Confidentiality may be granted for studies collecting information that, if disclosed, could have adverse consequences for participants, such as damage to their financial standing, employability, insurability, or reputation. By protecting researchers and institutions from being compelled to disclose information that would identify research participants, Certificates of Confidentiality help to minimize risks to subjects by adding an additional level of protection for maintaining confidentiality of private information. The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects. The Certificate of Confidentiality will also not be used to prevent disclosure to state or local authorities of events that the researchers are obligated to report, such as if research staff have strong reason to believe you are abusing a child or an elderly person, or if you and/or your teen have made credible threats of violence to self or others. In these cases, researchers may report it to appropriate authorities.

#### D. HOW BEING IN THE STUDY CAN BENEFIT YOU

There is no direct benefit to you or your teen of participating in this study. A potential indirect benefit of being in the study is that you and your teen may learn new ways to communicate about your teen's whereabouts and/or behavior, and while you are in the study, you will have an additional way of supervising your teen. Another potential indirect benefit of participating in this study is knowing that you and/or your teen are contributing to the development of technology that may someday help teens with externalizing behaviors/conduct disorders, their parents/guardians, and service providers.

## E. COSTS

There are no costs to you or your teen for participating in this study.

## F. PAYMENT TO PARTICIPANTS

You and your teen will each receive compensation for the study assessments you complete and can earn bonuses for completing at least 3 (Bonus 1) and all 4 (Bonus 2) of the assessments. Parents/Guardians can earn up to \$240 and teens can earn up to \$140. Payments will be issued by

checks mailed to your address. Your teen's payment will be issued to you so that you may choose how he/she receives it.

| Pa | yment | for | com | pleted | assessi | nents | and | bonuses | are | as | follows. |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | , | | | | | | | | | | |

| Study Time | Parent/Guardian | Teen | Optional | Parent/Guardian | Teen |
|---|---|---|---|---|---|
| Point | Compensation | Compensation | Bonus | Compensation | Compensation |
| Baseline | \$30 | \$25 | Bonus 1<br>(3 of 4) | \$30 | \$20 |
| Week 4 | \$40 | \$25 | Bonus 2<br>(4 of 4) | \$30 | \$20 |
| Week 8 | \$50 | \$25 | | | |
| Week 12 | \$60 | \$25 | | | |

After you and your teen complete the study, you will be able to use iKinnect for 3 additional months. If you received the other app for use in the study, we will send you access to iKinnect upon your completion of the study.

## **G. ALTERNATIVES**

The alternative to participating in this study is not participating in the study.

Results of this research will be used for the purposes described in this study. This information may be published, but you and your teen will not be identified.

Information that is obtained as part of this research that can be identified with you and/or your teen will remain confidential to the extent possible within State and Federal law. The investigators associated with this study, the sponsor, and the institutional review board(s) overseeing this research will have access to identifying information.

You and your teen's participation in this study is voluntary. You and/or your teen may refuse to take part in or stop taking part in this study at any time. You and/or your teen should tell the research staff person conducting the study if you decide to do this. You/your teen's decision not to take part in the study will not affect your current or future medical care, any benefits to which you are entitled, or your teen's legal status within the justice system.

The investigators and/or sponsor may stop you and/or your teen's participation in this study at any time if they decide it is in your best interest. They may also do this if you do not follow the investigator's instructions.

#### H. CLINICAL TRIALS REGISTRY DATABANK

A description of this clinical trial will be available on www.ClinicalTrials.gov, as required by US Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## **Parent/Guardian Volunteers Statement**

- I have been given a chance to ask questions about this research study. I am satisfied with the answers I was given.
- If I have any more questions about my participation in this study, would like to withdraw from the study, or become distressed from being in the study, I may contact: Dr. Linda Dimeff: (206) 384-7371 | Dr. Cindy Schaeffer: (410) 706-6855 | Angela Kelley Brimer: (206) 717-5666
- If I have questions about my rights as a research participant or if I have questions, concerns or complaints about the research, I may contact: Behavioral Health Research Collective's Institutional Review Board Chair, Dr. Travis Osborne at 206-374-0109. This includes any questions about my rights as a research participant in this study.
- I have been given a copy of this form for my own records.
- I agree to participate in this study.

| PARENT/GUARDIAN: If <u>YOU</u> wish to participate, you should sign here: | |
|---|---|
| Signature of Participating Parent/Guardian | Date |
| Printed Name of Participating Parent/Guardian | |
| We will also collect your data from iKinnect, if you are randomized to use il study, please provide permission for us to use these data. | Kinnect. To participate in the |
| Consent to obtain data from iKinnect: I authorize Evidence-Based access and use the data collected within iKinnect during my/my teen' | |
| Sometimes, the parent who participates in the study does not have legal g cannot legally sign for the teen). If you are not the teen's legal guardian, pl guardian complete the rest of this consent. | |
| Consent for Other Parent: I consent for my youth to participate with a different parent/caregiver in the day-to-day use of the research app and completion of the assessments as a part of this research study. | |
| LEGAL PARENT/GUARDIAN: If you wish for YOUR TEEN to participate, y | you should sign here: |
| I agree for my teen to participate in this study. | |
| Signature of Teen's Legal Parent/Guardian (Consent for Youth) | Date |
| We will also collect your teen's data from iKinnect, if your teen is randomiz participate in the study, please provide permission for us to use these data | |
| Consent to obtain data from iKinnect: I authorize Evidence-Based access and use the data collected within iKinnect during my/my teen' | |

## **Youth Volunteers Statement**

- I have had this research study explained to me and have been given a chance to ask questions about the study. I am satisfied with the answers I was given.
- If I have any more questions about my participation in this study, would like to withdraw from the study, or become distressed from being in the study, I may contact: Dr. Linda Dimeff: (206) 384-7371 | Dr. Cindy Schaeffer: (410) 706-6855 | Angela Kelley Brimer: (206) 717-5666
- If I have questions about my rights as a research participant or if I have questions, concerns or complaints about the research, I may contact: Behavioral Health Research Collective's Institutional Review Board Chair, Dr. Travis Osborne at 206-374-0109. This includes any questions about my rights as a research participant in this study.
- I agree to participate in this study.

| YOUTH: If you wish to pa | articipate, you should sign here: | |
|---------------------------|-----------------------------------|------|
| Signature of Youth Assent | | Date |
| Printed Name of Youth | | |
| Youth Age | Youth Date of Birth | |

## iKinnect Clinical Trial

## Evidence-Based Practice Institute, LLC CONSENT TO PARTICIPATE IN RESEARCH – Adult Youth Version

TITLE: Developing Mobile Technology to Enhance Multisystemic Therapy (MST)

Outcomes

**SPONSOR &** National Institute of Mental Health

PROTOCOL NUMBER: R44MH097349-A1

PRINCIPAL Linda Dimeff, PhD INVESTIGATORS: (206) 384-7371

Cindy Schaeffer, PhD (410) 706-6855

SITE: Evidence-Based Practice Institute, LLC

3303 South Irving Street Seattle, Washington 98144

**United States** 

OTHER STUDY-RELATED Julie Chung

PHONE NUMBER: Study Coordinator

(206) 717-5666

## This consent form contains important information to help you decide whether to participate in a research study.

- > Being in a study is voluntary your choice.
- If you join this study, you can still stop at any time.
- No one can promise that a study will help you.
- > Do not join this study unless all of your questions are answered.

## After reading and discussing the information in this consent form you should know:

- Why this research study is being done;
- What will happen during the study;
- Any possible benefits to you;
- The possible risks to you;
- Other options you could choose instead of being in this study;
- How your personal health information will be treated during the study and after the study is over;
- Whether being in this study could involve any cost to you; and
- What to do if you have problems or questions about this study.

## Please read this consent form carefully.

## A. PURPOSE & BACKGROUND

We have developed iKinnect, a new mobile app for teens who have behaviors like skipping school, physical fights, illegal behaviors, and arrests and their parents/guardians. iKinnect is designed to give teens rewards (like Google Play/Apple Store credit) for positive behavior, help parents/guardians and teens work together to meet behavior goals, and monitor teen activities and whereabouts. Right now, we are looking for parents/guardians and teens to use the app for 12 weeks (3 months) in real life and tell us their likes and dislikes as they use it. We will also ask that parents/guardians and teens complete phone interviews and online surveys at the start of the study (baseline) and at 4, 8, and 12 weeks.

You and your parent/guardian are being asked to volunteer for this research study. Your participation is completely voluntary (your choice). You do not have to be in this study if you do not want to. Parents/Guardians and teens are required to participate together as a pair. This means that both you and your parent/guardian must agree to participate in the study in order to enroll in it. Parents/Guardians and teens will participate together and pairs will be randomly assigned (like flipping a coin) to use either the iKinnect app or another app, called Life360, on your Android or Apple smartphones. All study interviews and surveys will be completed independently (on your own). We will want to talk with you and your parent/guardian about your views and opinions about how the app you were assigned to use is working for your family, what you like and dislike, and your suggestions for how to make it better. We will also ask about and evaluate the app's helpfulness/usefulness, how often you and your parent/guardian use the app, barriers you might experience to using the app, parenting practices, life stress, clarity of expectations, youth delinquent/prosocial behaviors, and motivation.

Finally, if you and your parent/guardian are assigned to use the iKinnect app, we will ask permission to talk with your service provider (case manager, therapist, etc.) at 8 weeks. We will ask your provider their opinions about you and your parent/guardian's use of the app, and whether they believe the app was helpful to your progress.

## **B. STUDY PROCEDURES**

If you agree to be in this study, the following will happen:

- 1. You and your parent/guardians will be randomly assigned (like flipping a coin) as a pair to use either the iKinnect or Life360 app on your Android or Apple smartphones.
- 2. We will give you and your parent/guardian a link to the iKinnect mobile app or another app used in the study. We will then ask that you each install the app on your Android or Apple smartphones and set it up. We are here to help with this process if you need.
- 3. You will be asked to use the app for 12 weeks. You will not be required to use any particular feature of the app if there is a specific reason why you and/or your parent/quardian prefer not to.
- 4. If you are assigned to use the iKinnect app, the research team will be able to access the information collected through your use of the app. iKinnect data that we collect will be coded with your study ID number and combined with the other participants' data. We will use this information to determine how iKinnect is being used by the parents/guardians and teens in this study. You will not be asked about this information during the study interview or surveys.
- 5. If you are assigned to use the Life360 app, you will be required to provide the following permissions in order for it to work properly: 1) location; 2) phone permission to allow Life360 to connect your phone to a live representative and authenticate that you are the one calling them if you choose to use that feature; and 3) network to allow Life360 to send and receive location information to and from family members on your private map. Other information regarding their terms of use, privacy policy, and data retention policies can be found in your app store or on the Life360 website.
- 6. You and your parent/guardians will each be asked to complete 4 study assessments over your 12 weeks of being in the study. These assessments will take place at the start of your participation

(also called "baseline") and during weeks 4, 8, and 12. Each assessment will include an interview and a brief set of surveys online. We expect no interview to last longer than 30 minutes and the surveys no longer than 30 minutes. Each assessment will last about 1 hour total. The assessments will be scheduled at a time that is most convenient for you. We recommend ensuring you are in a quiet, private place during the assessments. We will want to talk with you about your views and opinions on how the app is working for your family, what you like and dislike, and your suggestions for how to make it better. We will also ask about and evaluate the app's helpfulness/usefulness, how often you and your parent/guardian use the app, barriers you might experience to using the app, parenting practices, life stress, clarity of expectations, youth delinquent/prosocial behaviors, and motivation.

- 7. You will receive compensation for the study assessments you complete and can earn bonuses for completing at least 3 (Bonus 1) and all 4 (Bonus 2) of the assessments. You can earn up to \$140 for completing this study.
- 8. You and your parent/guardian's names will not be associated with the answers you provide during the interviews or on surveys. You have the right to not answer a question or withdraw from the study for any reason at any time if you choose, without penalty. You may contact Dr. Dimeff or Dr. Schaeffer at any time if you have any concerns or are feeling discomfort due to study participation.

## C. RISKS/DISCOMFORTS

There are seven kinds of potential risks to you for participating in this study:

1. Potential embarrassment of sharing your opinions (likes and dislikes) of the app with us in an interview and/or feeling possible distress when answering survey questions about your behaviors and your parent/guardian's behaviors.

## To reduce the risk of embarrassment and/or distress of sharing your opinions and other study data with us:

- During the study interviews, we will talk only about the app itself and how teens, parents/guardians, and service providers might use it; discussions about personal or private matters will not be allowed.
- If at any time you feel uncomfortable or embarrassed, you are encouraged to tell us right away.
- If you would like, we will tell the investigators of your concerns, and she will contact you to talk about how best to address your concerns.
- To lessen the anxiety that assessment procedures can cause, we have purposely designed the
  procedure to allow you to complete the assessments in the comfort of your own home. We are
  also available to answer any questions you may have or provide any assistance you might need
  during the assessments.
- You are free to stop your participation in the study at any time or refuse to answer any question you are uncomfortable answering.
- 2. Possibility of experiencing distress if you and your parent/guardian disagree about how the app should be used.

## To reduce the possibility of you or your parent/guardian experiencing distress if you disagree about how the app should be used:

- Research staff, including staff who are clinical psychologists, will be available to talk with you if this occurs and you would like to speak with someone about it.
- If your distress level is high, you, your parent/guardian, or a research staff member can inform your service provider about the distress and your provider can help you.

- You are free to withdraw from the study at any time if you find that participation is too distressing.
- 3. Potential embarrassment when using the app in a public place or when around people who you may know or who may not know you are in a research study.

To reduce the risk of embarrassment when using the app in a public place or when around people who you may know or who may not know you are participating in a research study:

- You are encouraged to only use the app when it feels comfortable to do so.
- We will never require you to use the app in a place or at a time when you do not want to use it.
- The server that houses the app is as resistant to hacking as possible; the protections for the server are similar to those used in banking or other commercial websites. This will help protect your information stored in the app, such as if the app server were "hacked" or if you or your parent/guardian were to lose your phone.
- As an added protection, all app-generated information will be stored on the server without your name. In addition, the app will only store data on the server, not on the phone itself.
- Using the app requires a login, and you can log out of the app at any time.
- Finally, as an added safeguard, we recommend you password-protect your smartphones (such as using a pin to unlock the phone) while you are in this study.
- 4. Possibility of incurring data charges while using the app.

## To avoid the possibility of incurring data charges while using the app:

- Check with your smartphone's data provider to ensure you know how much data you are allowed to use each billing period without incurring extra charges.
- Use the app only when on a Wi-Fi connection.
- If needed, log out of the app and only log back in when you are comfortable doing so.
- 5. Possible loss of confidentiality and security of your data.

To minimize risks to confidentiality associated with management and storage of data, including identification of participants who took part in this study or information collected about you while using the app, we will:

- Train and supervise research staff to ensure strict compliance with the data protection plan.
- Your answers during the interviews and on the surveys will be stored on a secure, passwordprotected drive accessible only to research staff.
- Your responses will be stored using a study ID number and the last four digits of your mobile
  device number. The list linking your name to the ID assigned to your information will be
  maintained in a separate, secured location, also password protected and accessible only to the
  research staff, and will be destroyed within three years from the date of collection.
- The information we collect from you will be associated only with your study ID number and the last four digits of your mobile device number, not your name, so nobody can identify it as yours. This is called "de-identified data." De-identified data will be kept indefinitely on the secure drive.
- 6. You could feel coerced (pressured) to participate.

## To minimize the risk that you will feel pressure or coercion to participate:

 You are under no obligation to participate in the study at all. You may stop your participation in the study at any time.

- To ensure that participation is indeed completely voluntary, we have informed your agency staff, including your service provider, on multiple occasions that participation in this study is and must remain completely voluntary (your choice).
- We will ask you and your parent/guardian separately for consent/assent to participate and inform each of you independently that being in the study is completely voluntary.
- You may refuse participation in any part of the study. You may also discontinue your
  participation in this study at any time, without in any way jeopardizing your treatment or legal
  status.
- 7. The final risk involves privacy and the protection of your data.

## To help us protect your privacy and data we collect during the study:

We have obtained a Certificate of Confidentiality from the National Institutes of Health. This Certificate helps protect your identifiable research information from forced or compelled disclosure. A Certificate of Confidentiality allows the investigator and others who have access to research records to refuse to disclose identifying information on research participants in civil, criminal, administrative, legislative, or other proceedings, whether federal, state, or local. The researchers will use the Certificate to resist any demands for information that would identify you. Certificates of Confidentiality may be granted for studies collecting information that, if disclosed, could have adverse consequences for participants, such as damage to their financial standing, employability, insurability, or reputation. By protecting researchers and institutions from being compelled to disclose information that would identify research participants, Certificates of Confidentiality help to minimize risks to subjects by adding an additional level of protection for maintaining confidentiality of private information. The Certificate cannot be used to resist a demand for information from personnel of the United States federal or state government agency sponsoring the project and that will be used for auditing or program evaluation of agency funded projects. The Certificate of Confidentiality will also not be used to prevent disclosure to state or local authorities of events that the researchers are obligated to report, such as if research staff have strong reason to believe you are abusing a child or an elderly person, or if you and/or your teen have made credible threats of violence to self or others. In these cases, researchers may report it to appropriate authorities.

## D. HOW BEING IN THE STUDY CAN BENEFIT YOU

There is no direct benefit to you of participating in this study. A potential indirect benefit of being in the study is that you may learn new ways to communicate about your whereabouts and/or behavior with your parent/guardian. Another potential indirect benefit of participating in this study is knowing that you are contributing to the development of technology that may someday help teens with externalizing behaviors/conduct disorders, their parents/guardians, and service providers.

## E. COSTS

There are no costs to you for participating in this study.

#### F. PAYMENT TO PARTICIPANTS

You and your parent/guardian will each receive compensation for the study assessments you complete and can earn bonuses for completing at least 3 (Bonus 1) and all 4 (Bonus 2) of the assessments. You can earn up to \$140. Payments will be issued by checks mailed to your parent/guardian. Your payment will be issued to your parent/guardian so that you may choose together how you receive it.

Your payment for completed assessments and bonuses are as follows.

| Study Time | Youth | Optional | Youth |
|------------|--------------|---------------------|--------------|
| Point | Compensation | Bonus | Compensation |
| Baseline | \$25 | Bonus 1<br>(3 of 4) | \$20 |
| Week 4 | \$25 | Bonus 2<br>(4 of 4) | \$20 |
| Week 8 | \$25 | | |
| Week 12 | \$25 | | |

After you and your parent/guardian complete the study, you will be able to use iKinnect for 3 additional months. If you received the other app for use in the study, we will send you access to iKinnect upon your completion of the study.

#### **G. ALTERNATIVES**

The alternative to participating in this study is not participating in the study.

Results of this research will be used for the purposes described in this study. This information may be published, but you will not be identified.

Information that is obtained as part of this research that can be identified with you will remain confidential to the extent possible within State and Federal law. The investigators associated with this study, the sponsor, and the institutional review board(s) overseeing this research will have access to identifying information.

Your participation in this study is voluntary. You may refuse to take part in or stop taking part in this study at any time. You should tell the research staff person conducting the study if you decide to do this. Your decision not to take part in the study will not affect your current or future medical care, any benefits to which you are entitled, or your legal status within the justice system.

The investigators and/or sponsor may stop your participation in this study at any time if they decide it is in your best interest. They may also do this if you do not follow the investigator's instructions.

#### H. CLINICAL TRIALS REGISTRY DATABANK

A description of this clinical trial will be available on www.ClinicalTrials.gov, as required by US Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## **Adult Youth Volunteers Statement**

- I have been given a chance to ask questions about this research study. I am satisfied with the answers I was given.
- If I have any more questions about my participation in this study, would like to withdraw from the study, or become distressed from being in the study, I may contact: Dr. Linda Dimeff: (206) 384-7371 | Dr. Cindy Schaeffer: (410) 706-6855 | Angela Kelley Brimer: (206) 717-5666
- If I have questions about my rights as a research participant or if I have questions, concerns or complaints about the research, I may contact: Behavioral Health Research Collective's Institutional Review Board Chair, Dr. Travis Osborne at 206-374-0109. This includes any questions about my rights as a research participant in this study.
- I have been given a copy of this form for my own records.
- I agree to participate in this study.

| We will collect your data from iKinnect. To participate in the study, please use this data. | provide permission for us to |
|---|---|
| Consent to obtain data from iKinnect: I authorize Evidence-Based Practice Institute, LLC to access and use the data collected within iKinnect during my use of the app. | |
| If <u>YOU</u> wish to participate, you should sign here: | |
| Signature of Adult Youth Participant | Date |
| Printed Name | |